CLINICAL TRIAL: NCT06018090
Title: Microembolic Detection in Acute Ischemic Stroke Patients With Atrial Fibrillation and Outcome - A Prospective Multicenter Study With Transcranial Doppler
Brief Title: Microembolic Detection in Acute Ischemic Stroke Patients With Atrial Fibrillation and Outcome
Status: Completed | Type: Observational
Sponsor: Centro Hospitalar De São João, E.P.E. (Other)
Collaborators: University of Giessen (Other); University of Padova (Other); University of Ostrava (Other); Clinical Hospital Centre Zagreb (Other)
Responsible Party: Principal Investigator, Pedro Castro, Professor, Centro Hospitalar De São João, E.P.E.
Other Study IDs: 362/19
Record Dates: First submitted 2023-08-25; First posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Infarction, Brain; Embolism; Atrial Fibrillation
Keywords: Infarction; Embolism; Atrial Fibrillation; Ultrasound; Transcranial Doppler
MeSH Terms: conditions — Brain Infarction; Embolism; Atrial Fibrillation; Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute Ischemic Stroke Patients with Atrial Fibrillation
  Interventions: Other: The presence and rate of MES measured by TCD monitoring

INTERVENTIONS:
Other: The presence and rate of MES measured by TCD monitoring — TCD monitoring within 24 hours from the last known well time. Bilateral M1 segments of middle cerebral artery were insonated at a single depth with 2-MHz transducers secured by a probe-holder.

SUMMARY:
This multicenter international prospective cohort study will include patients with AIS with a known or newly diagnosed anticoagulant-naïve AF. All centers will use the same transcranial Doppler machine for one-hour monitoring with bilateral 2-MHz probes within 24 hours of symptom onset. Recordings will be analyzed for MES by a blinded central reader. The primary aim is to determine the proportion of patients with MES and the association of MES with functional outcomes assessed by a modified Rankin scale (mRS) score at 90 days.

ELIGIBILITY:
Inclusion Criteria:

* acute ischemic stroke admitted to the Stroke Unit, history of AF/flutter or a new diagnosis of AF at the stroke, and with a possibility to be monitored within 24 hours after symptom onset.

Exclusion Criteria:

* use of anticoagulants at stroke onset; prosthetic valves; inadequate temporal bone window; uncooperative patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute ischemic stroke admitted to the Stroke Unit, history of AF/flutter, or a new diagnosis of AF at the time of stroke, and able possibility to be monitored within 24 hours after symptom onset.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-10-06 (Actual)

PRIMARY OUTCOMES:
Prevalence of MES | Within 24 hours of symptom onset
Poor functional outcome | 90-days after stroke

SECONDARY OUTCOMES:
Ordinal Shift Analysis of mRS scale score | 90-days after stroke

CONTACTS AND LOCATIONS:
Locations (1):
- Pedro Miguel Castro, Porto, Portugal

REFERENCES:
- [Derived] Castro P, Ferreira J, Malojcic B, Bazadona D, Baracchini C, Pieroni A, Skoloudik D, Azevedo E, Kaps M. Detection of microemboli in patients with acute ischaemic stroke and atrial fibrillation suggests poor functional outcome. Eur Stroke J. 2024 Jun;9(2):409-417. doi: 10.1177/23969873231220508. Epub 2023 Dec 27. PMID 38149620